CLINICAL TRIAL: NCT04116138
Title: Antisecretory Factor, Administered as an Enriched Egg Powder, Salovum®, as Supplementary Therapy for Primary Glioblastoma During Concomitant Radio-chemotherapy.
Brief Title: Antisecretory Factor in Primary Glioblastoma 1
Acronym: AFGBM1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peter Siesjö (Other)
Collaborators: Region Skane (Other); Lund University (Other); Skane University Hospital (Other); Lantmannen Medical AB (Other)
Responsible Party: Sponsor-Investigator, Peter Siesjö, Professor, Skane University Hospital
Organization: Skane University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFGBM1
Record Dates: First submitted 2019-09-26; First posted 2019-10-04 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2020-11

CONDITIONS: Glioblastoma; Cerebral Edema; Chemotherapy Effect
MeSH Terms: conditions — Glioblastoma; Brain Edema | interventions — antisecretory factor

STUDY DESIGN:
Intervention Model Description: Phase 1-2, open label, single arm, single center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Salovum (Experimental): Salovum®, an egg powder enriched for anti secretory factor.
  Interventions: Dietary Supplement: Salovum

INTERVENTIONS:
Dietary Supplement: Salovum — Egg yolk powder enriched for anti secretory factor
  Other Names: Antisecretory factor

SUMMARY:
This is a non-randomised, open-label, single center-centre, Phase I-II study in patients with newly diagnosed glioblastoma. 5 patients with newly diagnosed glioblastoma are enrolled in the study and will receive an egg powder enriched for antisecretory factor (AF), Salovum, daily from 2 days before concomitant radio-chemo therapy until 14 days after finalisation.The primary aim of the study is to asses safety and feasibility of this regimen.

DETAILED DESCRIPTION:
Glioblastoma (GBM) is the most common primary brain tumor and also has the worst prognosis with a mean survival time below 1 year and a 5-year survival rate of less than 2%.

AF is a 41kilodalton endogenous and essential protein encompassing antisecretory and anti-inflammatory effect. Endogenous AF activity increases after exposure to bacterial toxins and endogenous triggers of inflammation. The active amino-terminal portion of AF has been synthesized as a 16 amino acid peptide (AF-16) and has been used in animal experimental studies. Salovum® is a product based on egg yolk powder B221® and contains high levels of AF. Salovum® is classified as food for special medicinal purposes (FSMP) by the European Union.

Many tumors show elevated interstitial fluid pressure (IFP) compared to the surrounding tissue due to vascular leakage, providing a barrier for drug uptake in solid tumors, as well as poor perfusion, resulting in hypoxia and relative resistance to radiochemotherapy.

In a mouse model of malignant brain tumor, preliminary findings show that intratumoral infusion of AF-16 greatly enhances the effect of simultaneous intratumoral temozolomide treatment (90% and 40% survival, respectively). AF-16 also has preliminarily significant immune modulatory effects on myeloid cells in vitro, but also effects on the secretion of immune modulatory agents from tumor cells. AF-16 was reported to significantly reduce the IFP in xenotransplanted human glioblastoma by inhibiting an ionic pump, NKCC1, in the tumor tissue. Both Salovum® and AF-inducing specific processed cereals (SPC) prolonged survival in the same models. Systemic temozolomide treatment combined with AF inducing SPC completely blocked tumor growth in GBM xenografts. Likewise, SPC treatment abrogated 90% of pre-established syngeneic tumors in immune competent animals.

Mechanistically, it remains unclear whether AF's effect in tumor models is mediated through decrease of IFP and/or immunomodulation. Also, an effect on the complement system through modulation of circulating complement complexes with proteasome units has been proposed.

Salovum® has been administered to patients with various diseases as, inflammatory bowel disease, Mb Ménière and mastitis and traumatic brain injury without signs of any adverse effects.

The described study is a safety and feasibility study and if these criteria are fulfilled, will be followed by a randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Pathology verified glioblastoma
2. Age 18-69 years
3. Surgical treatment-biopsy or resection.
4. Scheduled full concomitant radiochemotherapy treatment with radiation (60 Gy) and temozolomide,
5. Informed consent

Exclusion Criteria:

1. No informed consent
2. Egg yolk allergy

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse | Cumulative from day 1 to 80
  Treatment related adverse events as assessed by CTCAE v 5.0
Number of participants with completion of prescribed Salovum treatment | Cumulative from day 1 to 80
  Defined as completing prescribed full Salovum treatment

SECONDARY OUTCOMES:
Number of participants with altered blood levels of triglycerides and cholesterol | Change from baseline at day 20, 57 and 70.
  Blood levels of triglyceride and cholesterol above normal range or increased from baseline
Number of participants with reduced or no steroid intake | Change from baseline at day 7, 14, 21, 28, 35, 42, 49, 56, 63 and 70.
  Intake of oral corticosteroids assessed weekly during and after intervention.
Number of participants with detetable blood levels antisecretory factor | Change from baseline at day 20, 57 and 70.
  Analysis of anti secretory factor-16 (AF-16) blood levels by enzyme linked immunoassay
Number of participants with altered blood levels of inflammatory cytokines | Change from baseline at day 20, 57 and 70.
  Analysis of interleukin-6 (IL-6), interleukin- (IL-8), monocyte chemotactic protein-1 (MCP-1), macrophage inflammatory protein-1a (MIP-1a), macrophage inflammatory protein-1b (MIP-1b) by multiplex analysis

OTHER OUTCOMES:
Cognitive function | Change from baseline at day 20, 57 and 70.
  Number of participants with decreased cognitive function assessed by Mini Mental State Examination (MMSE)
Number of participants with decreased neurological function | Change from baseline at day 20, 57 and 70.
  Neurologic function assessed by Neurologic Assessment in Neuro-Oncology (NANO) scale. Minimum 0 (no deficits) and maximum 25 (maximum deficits)
Number of participants with decreased performance | Change from baseline at day 20, 57 and 70.
  Number of participants with decreased performance assessed by Eastern Oncology Cooperative Group (ECOG) scale. Minum 0 (normal function) and maximum 4 (maximum disability)
Number of participants with decreased quality of life | Change from baseline at day 20, 57 and 70.
  Number of participants with decreased quality of life assessed by European Organization of Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) C30 and brain cancer module (BN20) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Peter Siesjö, MD, PhD, Principal Investigator — Skane University Hospital
Locations (1):
- Department of Neurosurgery, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
As there are only 5 patients in this study individual patient data without age and gender will be shared after publication
Supporting Information: Study Protocol
Time Frame: De identified individual patient data will be made available from 3 months after publication up to 24 months after publication
Access Criteria: By request from researcher

REFERENCES:
- [Derived] Ehinger E, Kopecky J, Darabi A, Visse E, Edvardsson C, Tomasevic G, Cederberg D, Belting M, Bengzon J, Siesjo P. Antisecretory factor is safe to use as add-on treatment in newly diagnosed glioblastoma. BMC Neurol. 2023 Feb 18;23(1):76. doi: 10.1186/s12883-023-03119-4. PMID 36803465